CLINICAL TRIAL: NCT04378322
Title: Sustainable Weight Loss Study: Nutrition Support Tools and Weight Loss Among Obese People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zipongo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 102
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Obesity
Keywords: weight loss; digital; nutrition; healthy eating; food purchasing; meal planning; obese; online; MyPlate
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nutrition and food purchasing tool + telenutrition (Active Comparator): Participants will use an online nutrition and food purchasing tool in addition to telenutrition.
  Interventions: Behavioral: Nutrition and food purchasing tool + telenutrition
- Nutrition and food purchasing tool (Active Comparator): Participants will use an online nutrition and food purchasing tool.
  Interventions: Behavioral: Nutrition and food purchasing tool
- Nutrition education tool (Active Comparator): Participants will be exposed to an online nutrition education materials.
  Interventions: Behavioral: Nutrition education tool

INTERVENTIONS:
Behavioral: Nutrition and food purchasing tool + telenutrition — Participants will be asked to use a meal planning and food purchasing feature regularly (at least once every two weeks) and schedule appointments with a registered dietitian.
  Arms: Nutrition and food purchasing tool + telenutrition
Behavioral: Nutrition and food purchasing tool — Participants will be asked to use a meal planning and food purchasing feature regularly (at least once every two weeks).
  Arms: Nutrition and food purchasing tool
Behavioral: Nutrition education tool — Participants will be asked to review nutrition education materials online.
  Arms: Nutrition education tool

SUMMARY:
The purpose of this research study is to determine the effectiveness of nutrition tools to support weight loss among obese individuals. All participation will be based online and there will be no in-person visits. Participants will be given nutrition support tools for 6 months. Participants will be asked to report their weight and diet at the start of the study, and every month for 6 months during the study period. Participants will additionally be asked to report weight and diet at 12 months, 18 months, and 24 months after the start of the study. Total study duration will be 2 years.

DETAILED DESCRIPTION:
Obesity is a major public health burden. Weight loss among obese participants may improve future health outcomes and financial burden to the healthcare system and employers.

The effect of personalized meal planning and online food purchasing and delivery on weight loss and management is unknown.

Design: This trial is an online, three-arm randomized trial to compare a meal planning and telenutrition tool, a meal planning tool only, and MyPlate optimization.

Participants will be assigned to randomly assigned in a 1:1:1 ratio to one of the three groups.

Participants will follow the intervention for 6 months after randomization and will be followed for an additional 1.5 years after randomization.

Participants will report dietary behavior and weight at baseline and each month of the intervention (6 months), 12 months, 18 months, and 24 months.

Population Approximately 300 participants will be enrolled and randomized (100 per arm). Participants will be adults living in New York state who are obese (at least a BMI of 30 kg/m2).

Outcomes Primary outcome: weight change after 6 months Other outcomes: waist circumference; blood pressure, dietary changes, cooking, meal planning, and eating out frequencies

ELIGIBILITY:
Inclusion Criteria:

BMI ≥ 30 kg/m2 Male or female 18 or older Non-institutionalized Able and willing to provide informed consent Willing to change diet for 3 months Has access to a scale to weigh themselves Lives in NY state

Exclusion Criteria:

Refuse or are unable to provide informed consent to participate in the study Undergoing active cancer treatment Has type 1 or 2 diabetes Stage 3+ CKD or kidney failure Are pregnant or breastfeeding, have given birth in the last three months, or are planning to be pregnant in the next 3 months Report of congestive heart failure Diagnosed with an eating disorder (e.g. anorexia nervosa or bulimia nervosa) Current or former Zipongo users

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-05-04 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Weight change | Baseline and end of months 1, 2, 3, 4, 5, 6, 12, 18, and 24
  Weight will be measured using a scale and self-reported.

SECONDARY OUTCOMES:
Waist circumference | Baseline and end of months 1, 2, 3, 4, 5, 6, 12, 18, and 24
  Waist circumference will be measured using a tape measure and self-reported.
Blood pressure | Baseline and end of months 1, 2, 3, 4, 5, 6, 12, 18, and 24
  Blood pressure will be a self-reported assessment at a clinic or pharmacy.
Change in diet quality | Baseline and end of months 1, 2, 3, 4, 5, 6, 12, 18, and 24
  Diet quality will be assessed using a food frequency questionnaire.

IPD SHARING:
Plan to Share IPD: No